CLINICAL TRIAL: NCT02313506
Title: Feasibility and Preliminary Efficacy of an Activity Tracker-driven Intervention for Promoting Physical Activity in People Living With Osteoarthritis of the Knee
Brief Title: Feasibility of a Wearable-enabled Intervention for Promoting Physical Activity in People Knee OA
Acronym: TRACK-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Arthritis Research Centre of Canada (Other); Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H14-02631
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-09

CONDITIONS: Knee Osteoarthritis; Joint Diseases
Keywords: Physical activity; Exercise; Osteoarthritis; Knee; Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Motor Activity; Osteoarthritis; Arthritis

STUDY DESIGN:
Intervention Model Description: This study used a delayed control design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Active Comparator): Education session, Fitbit Flex, and remote coaching by a PT. These three components of the intervention will be delivered to the participants in Month 1. At the end of the education session, the PT will help participants set personal activity goals. In Month 1, participants will use the Fitbit Flex. The PT will review the progress with participants via 20-minute weekly phone calls and progressively modify their activities. In Month 2, they will continue using the Fitbit and have access to a PT via email as needed, but no weekly phone calls.
  Interventions: Behavioral: Education session, Fitbit Flex, and remote coaching by a PT
- Delayed Intervention Group (Placebo Comparator): Same intervention with a 1 month delay: The full intervention will be initiated in Month 2 with a brief education session, use of Fitbit Flex, and counselling by a physiotherapist. The trial will conclude at the end of Month 2.
  Interventions: Behavioral: Same intervention with a 1 month delay

INTERVENTIONS:
Behavioral: Education session, Fitbit Flex, and remote coaching by a PT — Participants will receive a brief education session, use of a commercially available physical activity tracker (Fitbit Flex), and remote counselling by a PT. Intervention will be received immediately.
  Arms: Immediate Intervention Group
Behavioral: Same intervention with a 1 month delay — The Delayed Intervention Group will receive the same intervention as the Immediate Intervention Group, but with a 1 Month delay.
  Arms: Delayed Intervention Group

SUMMARY:
Physical activity is an essential first-line treatment for patients with knee osteoarthritis (OA). However, a 2013 systematic review found only 13% met the activity recommendation of 150 minutes or more per week. The primary goal of this pilot randomized controlled trail is to assess the feasibility and preliminary efficacy of a multi-component intervention/model of care involving a group education session, use of the Fitbit Flex (a wireless physical activity tracking device), and weekly telephone counselling by a physiotherapist (PT) to improve physical activity and reduce sedentary time in patients with knee OA.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is common (affecting 1 in 10), painful, and debilitating. Being physically active improves pain, mobility and quality of life for people living with knee OA; however, less than half of patients are active. Combining the best evidence in OA care and digital technology, the investigators propose a new model of care for improving physical activity in patients with OA.

The investigators primary objective is to determine the feasibility and preliminary efficacy of a multi-component model of care involving 1) a group education and structured goal-setting session, 2) the use of Fitbit Flex (a commercially available physical activity tracker) and 3) weekly telephone activity counselling by a physiotherapist for improving physical activity and reducing sedentary time in patients with knee OA.

In this pilot randomized controlled trial the investigators hypothesize that compared to a control group (i.e. the Delayed Intervention group), participants in the Immediate Intervention Group will 1) increase moderate/vigorous physical activity (MVPA), 2) reduce sedentary time, 3) improve OA disease status, and 4) improve abilities to self-manage their condition.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician confirmed diagnosis of knee osteoarthritis OR are both 1) over 50, and 2) have experienced 4 weeks of pain, aching, or discomfort in or around the knee during the last year (equal to or more than 28 separate or consecutive days).
* Have no previous diagnosis of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, polymyalgia rheumatica, connective tissue diseases, fibromyalgia or gout.
* Have no history of using disease-modifying anti-rheumatic drugs or gout medications.
* Have no prior knee replacement surgery, and not on a waiting list for total knee replacement surgery.
* Have no history of acute injury to the knee in the past 6 months.
* Have not had surgery in the back, hip, knee, foot or ankle joints in the past 12 months.
* Have an email address and daily access to a computer with internet connection.
* Be able to attend a 2-hour education session at the Mary Pack Arthritis Centre.

Exclusion Criteria:

* Have a body mass index of equal to or greater than 40
* Have received a steroid injection in a knee in the last 6 months
* Have received a hyaluronate injection in a knee in the last 6 months
* Use medication that may impair activity tolerance (e.g. beta blockers)
* Are at risk when exercising, as identified by the Physical Activity Readiness Questionnaire (PAR-Q)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PT, PhD, Principal Investigator — Arthritis Research Canada; University of British Columbia
Locations (1):
- Arthritis Research Canada, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li LC, Sayre EC, Xie H, Clayton C, Feehan LM. A Community-Based Physical Activity Counselling Program for People With Knee Osteoarthritis: Feasibility and Preliminary Efficacy of the Track-OA Study. JMIR Mhealth Uhealth. 2017 Jun 26;5(6):e86. doi: 10.2196/mhealth.7863. PMID 28652228
- [Derived] Clayton C, Feehan L, Goldsmith CH, Miller WC, Grewal N, Ye J, Yoo JY, Li LC. Feasibility and preliminary efficacy of a physical activity counseling intervention using Fitbit in people with knee osteoarthritis: the TRACK-OA study protocol. Pilot Feasibility Stud. 2015 Aug 22;1:30. doi: 10.1186/s40814-015-0027-x. eCollection 2015. PMID 27965808
- See also: Study webpage — http://arthritis.rehab.med.ubc.ca/2015/02/04/improving-physical-activity-using-a-wearable-activity-tracker-pilot-testing-a-new-model-of-care-for-knee-osteoarthritis-track-oa/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our recruitment strategy identified 46 eligible individuals. Recruitment was from January 2015 to March 2015. Participants were recruited from 1) postings on Facebook, Twitter, Kajiji, Craigslist, and the Arthritis Research Canada website, 2) emails sent by the Arthritis Consumer Experts the Vancouver Coastal Health Research Institute to its staff.
Period: Overall Study
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Group | Delayed Intervention Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (9.7) | 58.7 (6.0) | 55.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 17 | 17 | 34
Marital Status [Count of Participants; unit: Participants]
  Married/Common Law | 11 | 14 | 25
  Separated/ Divorced | 4 | 1 | 5
  Widowed/ Never Married/ Other | 2 | 2 | 4
Gross annual household income [Count of Participants; unit: Participants]
  Under $12,000 | 1 | 1 | 2
  $12,001 - $24,000 | 0 | 1 | 1
  $24,001 - $40,000 | 0 | 2 | 2
  $40,001 - $60,000 | 4 | 1 | 5
  $60,001 - $80,000 | 0 | 0 | 0
  $80,001 - $100,000 | 2 | 1 | 3
  Over $100,000 | 7 | 7 | 14
  No answer | 3 | 4 | 7
Diagnosed with OA [Count of Participants; unit: Participants]
  Yes | 11 | 9 | 20
  No, but met the 'likely OA' criteria | 6 | 8 | 14
In general, would you say your health is ... [Count of Participants; unit: Participants]
  Excellent | 5 | 1 | 6
  Very good | 5 | 6 | 11
  Good | 4 | 9 | 13
  Fair | 3 | 1 | 4
  Poor | 0 | 0 | 0
Compared to one year ago, how would you rate your health in general? [Count of Participants; unit: Participants]
  Much better | 1 | 0 | 1
  Somewhat better | 0 | 1 | 1
  About the same | 15 | 12 | 27
  Somewhat worse | 1 | 4 | 5
  Much worse | 0 | 0 | 0
Comorbid conditions [Median (Inter-Quartile Range); unit: comorbid conditions] | 3 [2 to 4] | 2 [2 to 3] | 2.5 [2 to 4]
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (4.5) | 25.4 (4.2) | 27.2 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Moderate-to-Vigorous Physical Activity (MVPA)
Description: Participants wore a SenseWear Mini device for 7 days at baseline, and Months 1 and 2. We calculated the average time spent in MVPA accumulated in bouts per day. A bout is defined as 10 consecutive minutes or more at the level of 3 or higher METs, with allowance for interruption of up to 1 minute below the threshold.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: Minutes per day
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
Minutes per day
  Baseline | 41.3 (51.6) | 66.5 (71.0)
  1 Month | 64.2 (70.5) | 56.0 (60.1)
  2 Months | 67.7 (85.8) | 81.9 (64.4)
Statistical Analysis 1: Comparison: Immediate Intervention Group vs Delayed Intervention Group; ANCOVA was performed to evaluate the effect of the group type on the outcome measures after adjusting for blocking and baseline (T0). We assessed 3 planned contrasts of changes in outcome measures over time. Contrast 1 compared T0-T1 between the 2 groups to determine if the intervention was superior to the control; Test type: Superiority; p = 0.02, ANCOVA — No adjustment was made for multiple comparisons because Type II error is a greater concern than Type I error in feasibility studies; Mean Difference (Net) = -31.1, 95% CI 2-sided [-56.6 to -5.7]
Statistical Analysis 2: Comparison: Immediate Intervention Group vs Delayed Intervention Group; ANCOVA was performed to evaluate the effect of the group type on the outcome measures after adjusting for blocking and baseline (T0). We assessed 3 planned contrasts of changes in outcome measures over time. Contrast 2 compared T0-T1 in the immediate group against T1-T2 in the delayed group; Test type: Superiority; p = 0.71, ANCOVA; Mean Difference (Net) = 4.6, 95% CI 2-sided [-19.6 to 28.9]
Statistical Analysis 3: Comparison: Immediate Intervention Group vs Delayed Intervention Group; ANCOVA was performed to evaluate the effect of the group type on the outcome measures after adjusting for blocking and baseline (T0). We assessed 3 planned contrasts of changes in outcome measures over time. Contrast 3 compared T0-T1 in the immediate group against T0-T2 in the delayed group; Test type: Superiority; p = 0.29, ANCOVA; Mean Difference (Net) = -11.0, 95% CI 2-sided [-31.1 to 9.1]

2. Secondary Outcome: Time Spent in Sedentary Behavior
Description: We calculated the average daily time spent with an energy expenditure of 1.5 METs or lower, occurring in bouts of > 20 minutes during waking hours.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: Minutes per day
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
Minutes per day
  Baseline | 548.4 (169.1) | 453.3 (180.5)
  1 Month | 524.9 (192.1) | 492.8 (164.8)
  2 Months | 523.9 (200.2) | 393.1 (144.2)

3. Secondary Outcome: KOOS - Symptoms
Description: Symptoms were measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 70.6 (15.8) | 70.4 (14.9)
  1 Month | 68.3 (18.4) | 66.8 (18.2)
  2 Months | 72.5 (20.2) | 73.2 (15.4)

4. Secondary Outcome: KOOS - Pain
Description: Pain was measured by a Knee Injury and Osteoarthritis Outcome Score subscale. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 74.5 (16.2) | 68.6 (16.1)
  1 Month | 71.4 (17.5) | 71.6 (15.2)
  2 Months | 79.1 (13) | 74 (15.4)

5. Secondary Outcome: KOOS - Activities of Daily Living
Description: Activities of Daily Living was measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 81.8 (17.1) | 78.3 (15.9)
  1 Month | 75.1 (19.7) | 79.1 (18.9)
  2 Months | 83 (14.9) | 82.2 (17.1)

6. Secondary Outcome: KOOS - Sport and Recreation Function
Description: Sport and Recreation Function was measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 55.6 (29.5) | 51.2 (26.0)
  1 Month | 54.7 (28.3) | 54.4 (31.4)
  2 Months | 64.4 (28.4) | 55.6 (22.6)

7. Secondary Outcome: KOOS - Knee-related Quality of Life
Description: Quality of life was measured by Knee Injury and OA Outcome Score (KOOS). The KOOS measures knee osteoarthritis disease status and consists of five sub-scales: knee pain, stiffness, daily activity, sports/recreation, and quality of life. Scores range from 0 to 100, with higher being better.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 53.3 (18.4) | 47.4 (16.1)
  1 Month | 51.8 (19.5) | 48.9 (19.3)
  2 Months | 56.6 (20.2) | 52.3 (18)

8. Secondary Outcome: Partners in Health Scale
Description: The Partners in Health Scale is a 12-item measure designed to assess disease self-management abilities including knowledge of health conditions, ability to participate in decision-making with health care professionals, and ability to pursue a healthy lifestyle. Scores range from 0 to 96, with lower being better.
Time Frame: Baseline; 1 month and 2 months from baseline
Population: The number of participants analyzed is the same as the number of participants assigned to each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 17 | 17
score on a scale
  Baseline | 21.9 (17.6) | 26.8 (15.3)
  1 Month | 17.2 (17) | 31.9 (17.9)
  2 Months | 21.6 (21.9) | 22.9 (15.2)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked using a monthly log (self-reported) over the duration of the study (6 months) for each participant.
Description: We tracked self-reported adverse events (falls, cardiovascular and musculoskeletal events).
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Our sample was physically active at baseline. Also, the majority of our participants were women. Men and women may respond to behavioral interventions differently, but we are unable to examine the effect of sex on the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No